CLINICAL TRIAL: NCT03941587
Title: A Multi-center Randomized Clinical Trial Comparing Intravitreal Aflibercept Monotherapy vs Aflibercept Combined With Reduced Fluence PDT for the Treatment of Polypoidal Choroidal Vasculopathy
Brief Title: Comparing Intravitreal Aflibercept Monotherapy vs Aflibercept Combined With Reduced Fluence PDT in PCV Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: National University Hospital, Singapore (Other); Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Gemmy Cheung Chui Ming, Professor, Singapore National Eye Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R1735/58/2020
Record Dates: First submitted 2019-04-24; First posted 2019-05-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-12

CONDITIONS: Polypoidal Choroidal Vasculopathy
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — aflibercept; Verteporfin

STUDY DESIGN:
Intervention Model Description: Multi-center randomized, double-masked clinical trial.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aflibercept + RF-PDT (Active Comparator): Patients with symptomatic macular PCV (n=80) as confirmed by Indocyanine green Angiography(ICGA) will be treated with Aflibercept (dosage=2mg/0.05ml) through an intravitreal injection + RF-PDT ( 6mg/m2 intravenous infusion of Verteporfin followed by laser light at a dose rate of 25 Joules/cm2) at baseline.
  Aflibercept- 1st treatment (baseline) followed by minimum retreatment interval of 4 weeks (from Baseline to week 8) and then retreatment at intervals of 4 weeks pro re nata (PRN) retreatment( week 12-48). Primary endpoint at week 52.
  RF-PDT treatment at baseline followed by pro re nata (PRN) at 12 week intervals.
  At each visit, subjects will be assessed based on BCVA, ophthalmic examination and Optical Coherence Tomography (OCT)
  Interventions: Drug: Aflibercept + reduced fluence photodynamic therapy (RF-PDT)
- Aflibercept + sham RF-PDT (Active Comparator): Patients with symptomatic macular PCV (n=80) as confirmed by Indocyanine green Angiography(ICGA) will be treated with Aflibercept (dosage=2mg/0.05ml) through an intravitreal injection, at baseline. A minimum of 1 injection(baseline) followed by minimum pro re nata (PRN) retreatment interval of 4 weeks ( from baseline to week 8) and then a minimum of 4 weeks retreatment thereafter (week 12-48). Primary endpoint at week 52.
  Sham RF-PDT treatment at baseline followed by pro re nata (PRN) at 12 week intervals.
  At each visit, subjects will be assessed based on Best Corrected Visual Acuity (BCVA), ophthalmic examination and Optical Coherence Tomography (OCT)
  Interventions: Drug: Aflibercept + sham reduced fluence photodynamic therapy (RF-PDT)

INTERVENTIONS:
Drug: Aflibercept + reduced fluence photodynamic therapy (RF-PDT) — Aflibercept dosage of 2mg in 0.05ml along with intravenous infusion of Verteporfin (6mg/m2)followed by laser light at a dosage of 25Joule/cm2
  Other Names: Eylea; Visudyne
  Arms: Aflibercept + RF-PDT
Drug: Aflibercept + sham reduced fluence photodynamic therapy (RF-PDT) — Aflibercept dosage of 2mg in 0.05ml along with sham photodynamic therapy
  Other Names: Eylea
  Arms: Aflibercept + sham RF-PDT

SUMMARY:
In this study, we aim to evaluate the efficacy and safety of an individualized dosing schedule comprising Aflibercept and RF-PDT in patients with polypoidal choroidal vasculopathy (PCV). The primary objective is to compare the polyp closure rate at week 12 between the 2 treatment groups. The secondary aims include comparing visual, anatomical, treatment burden and clinical biomarkers between each treatment group.

DETAILED DESCRIPTION:
Age related macular degeneration (AMD) is one of the leading causes of blindness worldwide. In its exudative or wet form, choroidal neovascularization (CNV) causes an exudative maculopathy resulting in sudden loss of vision with severe effects on patients' quality of life. Intravitreal injections of anti-vascular endothelial growth factor agents (anti-VEGF) have become the mainstay of treatment for AMD CNV and has been shown to have favorable outcomes in most AMD CNV subtypes. In the Asian population, however, a particular subtype called polypoidal choroidal vasculopathy (PCV), which affects about 50% of exudative maculopathy, has been shown to have less favorable response to anti-VEGF therapy.

The best treatment option for PCV has remained unclear. Current best evidence is from 2 recent randomized controlled trials, the EVEREST II trial which compares the efficacy of ranibizumab with or without photodynamic therapy (PDT) for treatment of PCV and the PLANET trial which compares Aflibercept monotherapy against a rescue PDT when Aflibercept is deemed ineffective. Both trials have reported significant improvement in visual outcomes, however there remain significant unanswered questions and unmet needs regarding the use of Aflibercept and PDT as the best treatment for PCV.

In this study, we aim to compare the efficacy of combination Aflibercept with RF-PDT (at baseline) and Aflibercept monotherapy. This particular strategy has not been studies before and represents the amalgamation of unanswered questions from the best evidence to date for the treatment of PCV.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 50 years old at the time of informed consent.
* Provide written informed consent.
* Willingness and ability to comply with all scheduled visits and study procedures.
* Confirmed diagnosis of symptomatic macular PCV based ICGA.
* Activity of PCV confirmed by exudative activity involving the macula on OCT or Fluorescein Angiography (FA) or both.

  * Presence of intra retinal or subretinal fluid/blood as seen on OCT
  * Treatment naïve

    * NO previous treatment with intravitreal anti-VEGF agents, regardless of the indication
    * NO previous thermal laser in the macular region, or verteporfin photodynamic therapy (vPDT), regardless of indication
    * NO other previous treatment for neovascular AMD (nAMD), except oral supplements and traditional Chinese medicine
* An ETDRS BCVA of at least 4 letters (Snellen equivalent approximately 20/800 or better) in the study eye.
* Greatest Linear Dimension (GLD) of the total lesion area (BVN + polyps) <5400µm (~9 mucopolysaccharidoses (MPS) Disc Areas) as delineated by ICGA.

Exclusion Criteria: - Participant

* Medical condition that, in the opinion of the investigator, would preclude participation in the study (e.g. unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Participation in an investigational trial within 30 days of enrollment which involves treatment with unapproved investigational drug.
* Known allergy to any component of the study drug.
* Blood pressure> 180/110 (systolic above 180 OR diastolic above 110 on repeated measurements). If blood pressure is brought below 180/110 by anti-hypertensive treatment, individual can become eligible.
* Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization.
* Systemic anti-VEGF or pro-VEGF treatment within four months prior to randomization or anticipated use during the study.
* Amblyopia or blind in one eye Study Eye
* Eye with intra retinal or sub-retinal fluid due to other causes than PCV
* An ocular condition is present (other than PCV) that, in the opinion of the investigator, might affect intra or sub retinal fluid or alter visual acuity during the course of the study (e.g., Diabetic Macular Edema (DME), vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.)
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by more than three lines (i.e., cataract would be reducing acuity to worse than 20/40 if eye was otherwise normal).
* Any intraocular surgery within 1 month of enrollment
* Treatment with intra vitreal corticosteroids
* History of retinal detachment or surgery for retinal detachment
* History of vitrectomy
* History of macular hole
* Evidence of vitreomacular traction that may preclude resolution of macular edema > 4 disc areas of intra/sub retinal hemorrhage
* Aphakia
* Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis

Other Eye

* Active intraocular inflammation
* History of uveitis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Polyp Closure rate | 12 weeks
  polyp closure rate at week 12 between the 2 treatment groups.

SECONDARY OUTCOMES:
Optical Coherence Tomography | 12 months
  For evidence of intraretinal or subretinal fluid, ill-defined hyper-reflective material and/or new hemorrhage
Optical Coherence Tomography-Angiograph | 12 months
  For evidence of intraretinal or subretinal fluid, ill-defined hyper-reflective material and/or new hemorrhage
Color Fundus photography | baseline, month 3, month12
  inspect anomalies associated to diseases that affect the eye, and to monitor their progression
Autofluorescence Photography | baseline, month 3, month12
  Retinal imaging
Fundus Fluorescein Angiography | Baseline, month 3, month 12
  Retinal circulation
Intra Ocular Pressure (IOP) | Baseline, 12 months
  Fluid Pressure in eye

CONTACTS AND LOCATIONS:
Overall Officials: Gemmy Cheung Chui Ming, Principal Investigator — Singapore National Eye Centre
Locations (2):
- Singapore (2):
  - Singapore National Eye Centre, Singapore, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chong YJ, Teo KYC, Wong W, Tan ACS, Su X, Gilead N, Chan HH, Ibrahim F, Fenner B, Ong C, Sun C, Sim S, Chee C, Chakravarthy U, Cheung CMG. Aflibercept With vs Without Reduced-Fluence Photodynamic Therapy for Polypoidal Choroidal Vasculopathy: A Randomized Clinical Trial. JAMA Ophthalmol. 2025 May 1;143(5):393-399. doi: 10.1001/jamaophthalmol.2025.0250. PMID 40146166
- [Derived] Vyas CH, Cheung CMG, Tan C, Chee C, Wong K, Jordan-Yu JMN, Wong TY, Tan A, Fenner B, Sim S, Teo KYC. Multicentre, randomised clinical trial comparing intravitreal aflibercept monotherapy versus aflibercept combined with reduced-fluence photodynamic therapy (RF-PDT) for the treatment of polypoidal choroidal vasculopathy. BMJ Open. 2021 Jul 15;11(7):e050252. doi: 10.1136/bmjopen-2021-050252. PMID 34266844